CLINICAL TRIAL: NCT06590636
Title: Impact of Expressive Touching During Embryo Transfer on the Anxiety and Pregnancy Rate of Women Undergoing in Vitro Fertilization
Brief Title: Impact of Expressive Touching During Embryo Transfer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Duha Shaqalaih, PhD student, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1307/23
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: IVF-ET
Keywords: Embryo; Expressive Touching; Women; Pregnancy; Anxiety; In Vitro Fertilization
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infertile women (Experimental)
  Interventions: Procedure: Expressive touching
- Control group (No Intervention)

INTERVENTIONS:
Procedure: Expressive touching — Woman's anxiety level was measured with the State-Trait Anxiety Inventory scale Following these measurements, expressive touching that lasted 15-20 minutes was performed in the following manner.
  The hands of the expressive touching performer warmed to body temperature (should not be cold).
  The woman's hand close to the performer was placed between the hands of the expressive touching performer.
  The woman's palm was gently grasped with the palms of the expressive touching performer.
  The hand below was fixed and the upper part of the woman's hand was gently rubbed with the hand above.
  Before and after massaging, the woman's arms and shoulders were touched at intervals.
  During the procedure, the woman was called by her name, and verbal communication with the woman was continued by holding her hands firmly and sincerely as if a handshaking done.
  Before the woman's discharge from the center, her anxiety level was measured with the State-Trait Anxiety Inventory scale
  Arms: Infertile women

SUMMARY:
Infertile individuals report psychiatric symptoms and that their levels of anxiety and depression are significantly higher than in fertile controls .Thus,this study aimed to determine the effect of expressive touching during embryo transfer on the anxiety and pregnancy rate.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of primary infertility,
* Being over the age of 25 and under the age of 35
* Able to read and write Arabic,
* Women who will be applied assisted reproductive techniques such as IVF- ICSI-ET,
* Women with the same drugs and protocols used in IVF treatment was included in the study.

Exclusion Criteria:

* Women who have problems in understanding and perception,
* Having a diagnosis of secondary infertility wasn't included in the study

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
The State-Trait Anxiety Inventory Scale | Anxiety levels in women were measured using the State-Trait Anxiety Inventory (STAI) both before and after the embryo transfer procedure. The assessments were conducted within 5 to 10 minutes of each other to capture the immediate impact of the procedure
  The scale is a self-assessment questionnaire and, consists of 40 items rated on 4- point Likert scale. The scale consists of two sub-dimensions: the "state anxiety" has 20 items and is used to determine what is felt at a specific moment under certain conditions, and the "trait anxiety" has 20 items and is used to determine what has been felt in the last seven days. The scale includes reversed and non-reversed items. The score obtained from the reversed items is subtracted from the score obtained from the non-reversed items. Then, 50 points are added to this score for the state anxiety dimension and 35 points for the trait anxiety dimension, giving the total score. The score obtained from the two sub-dimensions ranges between 20 and 80. Higher scores indicate that the anxiety level is high

CONTACTS AND LOCATIONS:
Locations (1):
- Albasma a private IVF center, Gaza, Palestinian Territories

IPD SHARING:
Plan to Share IPD: No